CLINICAL TRIAL: NCT05118763
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, and Efficacy of Intranasal INNA-051 for Prevention of COVID-19 in Adults Following Close Contact With Individuals With SARS-CoV-2 Infection
Brief Title: Intranasal INNA-051 for Prevention of COVID-19 in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: ENA Respiratory Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INNA-051-COVID-PEP-01
Record Dates: First submitted 2021-10-27; First posted 2021-11-12 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — INNA-051

STUDY DESIGN:
Intervention Model Description: Randomised double blind placebo controlled parallel arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- INNA-051 arm 1 (Experimental): INNA-051 intranasal spray low dose administered once on each of Days 1, 4, 7 and 10
  Interventions: Drug: INNA-051
- INNA-051 arm 2 (Experimental): INNA-051 intranasal spray high dose administered once on each of Days 1, 4, 7 and 10
  Interventions: Drug: INNA-051
- Placebo (Placebo Comparator): Placebo intranasal spray high dose administered once on each of Days 1, 4, 7 and 10
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: INNA-051 — Liquid for intranasal administration
  Arms: INNA-051 arm 1; INNA-051 arm 2
Other: Placebo — Liquid for intranasal administration
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study of INNA-051 in adults following household contact with an individual with RT-PCR confirmed SARS CoV-2 infection. This study will evaluate 2 active dose levels of INNA-051 and placebo.

DETAILED DESCRIPTION:
Adults who have a household member with RT-PCR-confirmed SARS-CoV-2 infection and have been in close contact, and who test negative to SARS-CoV-2, will be randomized. Participants will receive 4 doses of study medication over a 10 day period, and complete symptoms scores and questionnaires. Development of COVID-19 symptoms will require collection of a nasal swab for RT-PCR testing.

Telephone visits will occur on Days 2, 4, 10, 21, 28, and 35. Additional visits will occur on Days 7, 14, and 42 (end of study).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent, provides signed written informed consent, and agrees to comply with protocol requirements.
2. Male or female aged ≥18 years.
3. Must have a symptomatic household contact ("index case") with rapid antigen/point of-care or RT-PCR-confirmed SARS-CoV-2 infection and onset of symptoms in the household contact within 5 days prior to screening.
4. Participants of non-childbearing potential. Non-childbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or vasectomy) or postmenopausal (amenorrhea for at least 12 months prior to screening without an alternative medical cause).

Exclusion Criteria:

1. Prior exposure to INNA-051.
2. Previous receipt of any full primary series SARS-CoV-2 vaccine or receipt of a booster vaccination following a full primary series within 12 months of screening.
3. Any symptoms of COVID-19 within 72 hours prior to screening. Symptoms may include fever (≥38°C), cough, sore throat, malaise, headache, muscle pain, nausea, vomiting, diarrhea, loss of taste and/or smell, shortness of breath, or difficulty breathing.
4. History of RT-PCR-confirmed SARS-CoV-2 infection within 6 months prior to screening.
5. Positive point-of-care rapid SARS-CoV-2 diagnostic test at the time of screening.
6. Body mass index ≥35 kg/m2.
7. History of human immunodeficiency virus, current chronic hepatitis B virus or hepatitis C virus infection or current tuberculosis.
8. History of chronic kidney disease (Stage 3 or higher).
9. Chronic lung disease (chronic obstructive pulmonary disease, moderate-to-severe poorly controlled asthma [as evident within the last month of awakening with asthma symptoms 1 or more times/week or use of short-acting beta-agonists 3 or more times/week], interstitial lung disease, cystic fibrosis, pulmonary hypertension).
10. History of significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis.
11. Current uncontrolled hypertension defined as average of 3 systolic blood pressure readings of ≥140 mmHg or an average of 3 diastolic blood pressure ≥90 mmHg.
12. History of chronic liver disease or documented evidence of liver fibrosis or cirrhosis.
13. History of hemoglobinopathy (sickle cell disease, thalassemia).
14. Chronic use of inhaled substances including tobacco, nicotine vapor, or cannabis (average of ≥5 cigarettes a day for ≥1 month within 1 year of screening or a 10 pack year history or equivalent).
15. History of neurological or neurodevelopmental conditions (e.g., Down's syndrome, dementia, migraine, epilepsy, stroke, seizure in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, or transverse myelitis).
16. History of malignancy in the last 5 years, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
17. History of immunodeficiency or chronic use (more than 14 continuous days) of any medication that may be associated with changes in the immune function including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs within 6 months of screening. Note: The use of low-dose topical and ophthalmic steroid preparations is permitted.
18. Use of nasal sprays (including but not limited to nasal glucocorticoids), intranasal washes, or other intranasal applications within 7 days prior to screening, or planned use during the study period.
19. Known allergy or sensitivity or contraindication to study drug or its excipients.
20. Treatment with any other investigational therapy or device within 30 days or within 5 half-lives, whichever is longer, prior to screening.
21. Female participants who are pregnant or trying to become pregnant, or who are breastfeeding.
22. Known history of substance abuse that in the investigator's judgment would prevent participant from providing informed consent or being able to comply with study procedures.
23. Other severe, acute, or chronic medical or psychiatric condition(s) that may increase the risk associated with study participation or interfere with the participant's ability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the ability of INNA-051 to reduce the incidence of symptomatic RT-PCR confirmed SARS-CoV-2 infection | To Day 14
  Incidence of symptomatic RT PCR confirmed SARS CoV 2 infection
Evaluate the safety and tolerability of INNA 051. | To Day 42
  Treatment emergent adverse events

SECONDARY OUTCOMES:
Evaluate the ability of INNA 051 to reduce the severity of symptoms in adults who develop RT PCR confirmed SARS CoV-2 infection after randomization | To Day 14 and to Day 28
  Incidences of RT PCR confirmed moderate or severe SARS-CoV-2 infection, or COVID 19 related death
Evaluate the ability of INNA 051 to reduce the severity of symptoms in adults who develop RT PCR confirmed SARS CoV-2 infection after randomization | To Day 14 and to Day 28
  Incidences of RT-PCR confirmed severe SARS-CoV-2 infection, or COVID-19-related death
Evaluate the ability of INNA 051 to reduce the severity of symptoms in adults who develop RT PCR confirmed SARS CoV-2 infection after randomization | On Day 14 and Day 28
  Modified FLU-PRO© total scores
Evaluate the ability of INNA 051 to reduce the severity of symptoms in adults who develop RT PCR confirmed SARS CoV-2 infection after randomization | On Day 14 and Day 28
  Modified FLU-PRO subscale scores for symptom severity by body system (nose, throat, eyes, chest/respiratory and gastrointestinal) in participants with RT PCR confirmed SARS CoV-2 infection
Evaluate the ability of INNA 051 to reduce the incidence of RT PCR confirmed SARS CoV-2 infection | To Day 28
  Incidence of symptomatic RT-PCR-confirmed SARS CoV-2 infection confirmed SARS CoV-2 infection
Evaluate the ability of INNA 051 to reduce the incidence of RT PCR confirmed SARS CoV-2 infection | To Day 14 and to Day 28
  Incidence of RT PCR confirmed SARS CoV-2 infection, through Day 14 and Day 28
Evaluate the ability of INNA 051 to reduce COVID 19 related healthcare utilization | To Day 14 and to Day 28
  Incidences of COVID 19 related emergency room visits, hospitalizations, or COVID 19 related death among participants with RT PCR confirmed SARS CoV-2 infection
Evaluate the ability of INNA 051 to reduce COVID 19 related healthcare utilization | To Day 14 and to Day 28
  2. Incidences of COVID 19 related medically attended visits (telemedicine, physician office, urgent care center, emergency room, hospitalization) or COVID 19 related death among participants with RT PCR-confirmed SARS CoV-2 infection

IPD SHARING:
Plan to Share IPD: No
No plan